CLINICAL TRIAL: NCT04973293
Title: The Safety and Feasibility of Preoperative Sintilimab Combined With Bevacizumab and Chemotherapy for Locally Advanced Resectable Non-Small Cell Lung Cancer
Brief Title: Preoperative Sintilimab Combined With Bevacizumab and Chemotherapy for Resectable Non-Small Cell Lung Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, Hecheng Li M.D., Ph.D, Professor, Ruijin Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RTS-014
Record Dates: First submitted 2021-07-13; First posted 2021-07-22 (Actual); Last update posted 2024-11-19 (Actual); Status verified 2024-11

CONDITIONS: Lung Neoplasm Malignant
Keywords: Non-small cell lung cancer; Neoadjuvant therapy; Immunotherapy
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — sintilimab; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Neoadjuvant treatment (Experimental): Participants will receive 4 doses of sintilimab (200 mg, IV) and bevacizumab (15 mg/kg, IV) every 3 weeks (Q3W). Participants will also receive 4 doses of carboplatin (AUC=5, IV) and pemetrexed (500 mg/m2, IV) Q3W.
  Surgery will be performed within 4 to 6 weeks after completion of preoperative therapy.
  After the second dose of sintilimab, bevacizumab and chemotherapy, contrast-enhanced chest CT will be performed. Patients with progression disease will receive surgery without the last 2 doses of treatment.
  Interventions: Drug: sintilimab; Drug: bevacizumab

INTERVENTIONS:
Drug: sintilimab — Sintilimab 200 mg, 4 cycles of treatment before surgery
  Other Names: IBI308; Xindili Dankang
Drug: bevacizumab — bevacizumab 15 mg/kg, 4 cycles of treatment before surgery
  Other Names: Bei Fa Zhu Dankang Zhusheye

SUMMARY:
Neoadjuvant chemotherapy followed by surgery has been recommended as the standard treatment for locally advanced and resectable non-small cell lung cancer (NSCLC). However, its efficacy remains to be improved. Drugs targeting PD-1/PD-L1 pathway have been proven to be effective for late-stage NSCLC, and anti-angiogenesis agents targeting VEGF (bevacizumab) has also been used for the first line treatment of advanced or metastatic NSCLC. Therefore, we conduct this single-arm clinical trial, which aims to investigate the safety and feasibility of neoadjuvant sintilimab combined with bevacizumab and chemotherapy followed by surgery in treating locally advanced and resectable NSCLC.

DETAILED DESCRIPTION:
Lung cancer is one of the most common malignancies around the world. Neoadjuvant chemotherapy followed by surgery has been recommended as the standard treatment for locally advanced and resectable non-small cell lung cancer (NSCLC). However, its efficacy remains to be improved. Bevacizumab targeting VEGF is a widely used antitumor drugs in different types of malignancies, including late-stage NSCLC. Immune checkpoint inhibitor (ICI) targeting PD-1 has also been confirmed to be effective in NSCLC patients. Therefore, we conduct this prospective single-arm clinical trial, to investigate the safety and feasibility of neoadjuvant sintilimab (ICI targeting PD-1) combined with bevacizumab and chemotherapy followed by surgery in treating locally advanced and resectable NSCLC. Twenty patients with stage II-IIIA NSCLC will be enrolled. And the primary endpoint of this study is the safety of this newly developed neoadjuvant treatment. The secondary endpoints are feasibility, radiological response and rate of major pathological response.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed, previously untreated and surgically resectable non-small cell lung cancer (stage II-IIIA, patients with squamous cell carcinoma or EGFR mutation should not be included);
2. Eastern Cooperative Oncology Group (ECOG) performance status 0-1;
3. Satisfactory preoperative laboratory testing and adequate pulmonary function for surgery;
4. Patients approve and sign the informed consent.

Exclusion Criteria:

1. Pancoast tumor, squamous cell carcinoma, large-cell carcinoma and sarcomatoid carcinoma;
2. Patients with active autoimmune disease or history of autoimmune disease;
3. Patients who have a condition requiring systemic treatment with either prednisone or other immunosuppressive medications;
4. Patients with a history of symptomatic interstitial lung disease;
5. History of allergy to study drug components;
6. Women must not be pregnant or breast-feeding;
7. Men with female partners that are not willing to use contraception;
8. Patients who have received prior chemotherapy, anti-angiogenesis therapy and immunotherapy for this malignancy or for any other past malignancy;
9. Patients who have received prior treatment for non-small cell lung cancer;
10. Any mental or psychological condition which would not permit the patient to complete the study or understand the patient information;
11. Patients who have major hemoptysis within the past 4 weeks, tumor has invasion or is close to great vessels;
12. Patients with high risk of major bleeding;
13. Patients who have arterial thrombotic events, esophageal varices, peptic ulcers, wounds or bone fractures;
14. Patients who have prior malignancies;
15. HIV, HBV, HCV infection or active pulmonary tuberculosis;
16. Underlying medical conditions that, in the Investigator's opinion, will make the administration of study drug hazardous or obscure the interpretation of toxicity or adverse events.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Safety (Rate of grade 3 and higher grade treatment-related adverse events) | From date of treatment allocation until surgery or up to at least 90 days after last dose of preoperative treatment
  Adverse events will be evaluated and recorded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (version 5.0).

SECONDARY OUTCOMES:
Feasibility (Completion rate of neoadjuvant treatment and surgery) | From date of treatment allocation until surgery, assessed up to 5 months
  Propotion of participants who complete neoadjuvant treatment and receive surgery within 42 days after preoperative therapies.
Major Pathological Response Rate | Two weeks after surgery
  Major pathologic response is predefined as no more than 10% of residual viable tumor cells in primary lesions.
Radiographic Response | From date of treatment allocation and during treatment period up to 4 months
  Radiographic response will be evaluated according to the Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1.

CONTACTS AND LOCATIONS:
Overall Officials: Hecheng Li, MD, PhD, Principal Investigator — Ruijin Hospital
Locations (1):
- Ruijin Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality, China